CLINICAL TRIAL: NCT02638701
Title: Infliximab Therapy for Dolichoectactic Vertebrobasilar Aneurysms
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Daniel L. Cooke, Assistant Professor of Radiology and Biomedical Imaging, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-16893
Record Dates: First submitted 2015-12-15; First posted 2015-12-23 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Aneurysm; Stroke; Vasculitis; Tumor Necrosis Factor-alpha
MeSH Terms: conditions — Aneurysm; Stroke; Vasculitis | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infliximab treatment (Experimental): Administer infliximab intravenously to patients with DVB aneurysms (3 mg/kg at 0, 3 and 7 weeks, then at 8-week intervals x 7) for a total of 12-months. Patients will undergo MR imaging at 0, 12, and 24-month time points.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Please see protocol for details.
  Other Names: Remicade

SUMMARY:
Patients harboring dolichoectactic vertebrobasilar (DVB) aneurysms are at risk of suffering SAH, ischemic stroke, and/or brainstem compression and many patients are not offered invasive treatment due to the futility of existing surgical methods. Consequently, there is demand for development of medical therapy for DVB aneurysms

DETAILED DESCRIPTION:
Dolichoectatic vertebrobasilar (DVB) aneurysms are fusiform in geometry and often large (< 10 cm) in size limiting traditional microsurgical clipping or endovascular coiling strategies. Collectively, DVB aneurysms represent ≤ 0.01% of all aneurysms (~ 600 US) and, consequently, their study is limited to a few small series. Despite their rarity, the location and geometry of DVB aneurysms make surgical intervention, microsurgical or endovascular, nearly uniformly fatal. Therefore, most DVB aneurysms are observed providing greater insight into their natural history than many more surgically amenable aneurysms. One series noted 28% of patients manifesting any neurological deficit, ischemic or hemorrhagic, over a 4 year interval with an overall mortality rate of ~ 20%.

Tumor necrosis alpha (TNFα). From the many implicated genetic pathways in aneurysm formation, tumor necrosis alpha (TNFα) has been noted a pivotal actor. In pre-clinical studies, the ability to inhibit TNFα induction prevents aneurysm rupture and even aneurysm growth altogether. In humans, TNFα inhibitor therapy has proven effective for many types of vascular inflammation including carotid wall thickening in the setting of rheumatoid arthritis. Over 12- and 24-month intervals, others have demonstrated significant decreases in carotid intima-media thickness in patients taking the TNFα inhibitor, infliximab. Furthermore, infliximab therapy has proven effective in refractory Kawasaki's disease, a condition characterized by post-infectious coronary artery inflammation in children. There is also evidence that infliximab therapy is effective in treatment of IVIG-refractory Kawasaki's disease including regressing coronary aneurysms. Despite the multitude of agents and indications both on and off-label, TNFα inhibitor therapy has not been used for the treatment of brain aneurysm.

ELIGIBILITY:
Inclusion Criteria:

1. Vertebral and/or basilar artery dolichoectactic aneurysm not amenable to microsurgical or endovascular treatment.
2. Age greater than 18 years at time of first study drug administration.

Exclusion Criteria:

1. Use of an anti-TNF or other biologic medication (Including but not limited to abatacept, rituximab, or tocilizumab) within the previous 12 months.
2. The following laboratory parameters at the Screening visit: Neutropenia (absolute neutrophil count < 1,500/microliter; Thrombocytopenia (platelets < 100,000/ • Anemia (hemoglobin < 8 g/dL); Greater than or equal to 3 times the upper limit of normal (ULN) for either of the following liver function tests (LFTs): aspartate transaminase (AST) or alanine transaminase (ALT); Renal insufficiency (serum creatinine> 2.0 mg/dL)
3. Purified protein derivative (PPD) test of > 5 mm induration regardless of prior BacilleCalmette Guerin vaccine administration or positive QuantiFERON®-TB Gold In-Tube Test (QFT-G_IT) without documentation of completed treatment or evidence of ongoing treatment of latent tuberculosis (TB) for 30 days. Subjects with active TB infection are excluded.
4. History of positive PPD, positive QuantiFERON®-TB Gold In-Tube Test (QFT-G_IT), or chest x-ray findings indicative of prior TB infection, without documentation of either treatment for TB infection or chemoprophylaxis for TB exposure
5. Presence of open leg ulcers
6. Chronic or persistent infection including but not limited to human immunodeficiency virus [HIV], untreated hepatitis B, listeriosis, TB, or other opportunistic infection). Patients with hepatitis C but without evidence of cirrhosis or significant hepatic dysfunction will be considered for inclusion on a case-by-case basis as will patients with chronic hepatitis B on anti-viral therapy.
7. Active infection or severe infections requiring hospitalization or treatment with intravenous (IV) antibiotics, IV antivirals, or IV antifungals within 30 days prior to randomization, or oral antibiotics, oral antivirals, or oral antifungals within 14 days prior to randomization
8. Receipt of a live vaccine within 4 weeks prior to randomization
9. History of malignancy within the past 5 years other than treated localized carcinoma in situ of the cervix or adequately treated non-metastatic squamous or basal cell skin carcinoma
10. Any medical condition, which, in the opinion of the investigator, would put the subject at risk by participation in the protocol
11. Women of childbearing potential who are sexually active and who do not agree to practice one of the following methods of contraception during the duration of the study: condoms, sponge, foams, jellies, diaphragm or intrauterine device; oral or parenteral contraceptives for 2 months prior to study product administration; a vasectomized partner; abstinence.
12. Pregnant (all women of childbearing potential must have a negative serum pregnancy test) or breastfeeding
13. Any investigational agent within the earlier of 4 weeks or 5 half-lives prior to randomization
14. History of drug or alcohol abuse within 6 months prior to randomization
15. Known allergy or hypersensitivity to any study products
16. Any psychiatric disorder that prevents the subject from providing informed consent
17. Inability or unwillingness to follow the protocol.
18. Unable to undergo MR imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in aneurysm volume (ml) | 12 months
  Our primary outcome for assessing the effectiveness of the infliximab treatment will be the reduction in aneurysm volume over the treatment course based on the 0 and 12 month MR scans. DVB aneurysm volume will be assessed by review of standardized 1.5 mm slices in the axial plane. The contour of the aneurysm using time-of-flight MR angiography sequences will generate a cross-sectional area at each slice level. The volume will be estimated by summing the imputed volume of each slice. Standard T1- and T2-weighted sequences will also be obtained, as well as iron-sensitive sequencing.

SECONDARY OUTCOMES:
Aneurysm computational fluid dynamic (CFD) metrics: flow velocity (ml/sec) | 12 months
  The investigators will capture MR-based, quantitative changes in the aneurysm computational fluid dynamics (CFD) metrics including flow velocity post 12-month IV infliximab administration. The investigators will compare pre- and post-treatment flow velocities using baseline and interval MR angiographic data. Such data is important in predication of aneurysm growth.
Aneurysm computational fluid dynamic (CFD) metrics: shear stress (pascal) | 12 months
  The investigators will capture MR-based, quantitative changes in the aneurysm computational fluid dynamics (CFD) metrics including wall shear stress post 12-month IV infliximab administration. The investigators will compare pre- and post-treatment CFD metrics using baseline and interval MR angiographic data. Such data is important in predication of aneurysm growth.
Aneurysm computational fluid dynamic (CFD) metrics: oscillatory index (0 - 0.5) | 12 months
  The investigators will capture MR-based, quantitative changes in the aneurysm computational fluid dynamics (CFD) metrics including oscillatory shear (OSI) index post 12-month IV infliximab administration. The investigators will compare pre- and post-treatment CFD metrics using baseline and interval MR angiographic data. Such data is important in predication of aneurysm growth. OSI ranges from 0 to 0.5, where 0 describes a total unidirectional WSS and the latter a purely unsteady, oscillatory shear flow with a net amount of zero WSS. Areas of high OSI are predisposed to endothelial dysfunction.
Aneurysm wall enhancement (ratio of signal post:signal pre contrast) | 12 months
  Continued improvements in higher field MR imaging have generated series noting the ability to not only resolve aneurysmal wall enhancement, but also the presence of such findings to reliably predict aneurysm growth and correlate with symptomatic events. To perform wall enhancement, the patient will first be scanned at 3T/7T using T1 weighted 3D black blood MRI technique (SPACE). Gadolinium will be injected and a 3D isotropic, high-resolution first-pass contrast-enhanced MR angiogram (CEMRA) will be obtained; immediately following that a post-contrast SPACE will be acquired. Contrast enhancement of the vessel wall will be graded as 0-2 scale or quantified by an enhancement ratio (Signal-post/Sigal-pre). Wall thickness can be estimated by the full width half maximal (FWHM) of the line profile across the vessel wall.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Cooke, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flemming KD, Wiebers DO, Brown RD Jr, Link MJ, Huston J 3rd, McClelland RL, Christianson TJ. The natural history of radiographically defined vertebrobasilar nonsaccular intracranial aneurysms. Cerebrovasc Dis. 2005;20(4):270-9. doi: 10.1159/000087710. Epub 2005 Aug 22. PMID 16123548
- [Background] Mangrum WI, Huston J 3rd, Link MJ, Wiebers DO, McClelland RL, Christianson TJ, Flemming KD. Enlarging vertebrobasilar nonsaccular intracranial aneurysms: frequency, predictors, and clinical outcome of growth. J Neurosurg. 2005 Jan;102(1):72-9. doi: 10.3171/jns.2005.102.1.0072. PMID 15658099
- [Background] Starke RM, Raper DM, Ding D, Chalouhi N, Owens GK, Hasan DM, Medel R, Dumont AS. Tumor necrosis factor-alpha modulates cerebral aneurysm formation and rupture. Transl Stroke Res. 2014 Apr;5(2):269-77. doi: 10.1007/s12975-013-0287-9. Epub 2013 Sep 20. PMID 24323710
- [Background] Ferrante A, Giardina AR, Ciccia F, Parrinello G, Licata G, Avellone G, Giardina E, Impastato R, Triolo G. Long-term anti-tumour necrosis factor therapy reverses the progression of carotid intima-media thickness in female patients with active rheumatoid arthritis. Rheumatol Int. 2009 Dec;30(2):193-8. doi: 10.1007/s00296-009-0935-2. PMID 19387646
- [Background] Del Porto F, Lagana B, Lai S, Nofroni I, Tinti F, Vitale M, Podesta E, Mitterhofer AP, D'Amelio R. Response to anti-tumour necrosis factor alpha blockade is associated with reduction of carotid intima-media thickness in patients with active rheumatoid arthritis. Rheumatology (Oxford). 2007 Jul;46(7):1111-5. doi: 10.1093/rheumatology/kem089. Epub 2007 Apr 20. PMID 17449484
- [Background] Burns JC, Best BM, Mejias A, Mahony L, Fixler DE, Jafri HS, Melish ME, Jackson MA, Asmar BI, Lang DJ, Connor JD, Capparelli EV, Keen ML, Mamun K, Keenan GF, Ramilo O. Infliximab treatment of intravenous immunoglobulin-resistant Kawasaki disease. J Pediatr. 2008 Dec;153(6):833-8. doi: 10.1016/j.jpeds.2008.06.011. Epub 2008 Jul 30. PMID 18672254
- [Background] Hasan DM, Chalouhi N, Jabbour P, Magnotta VA, Kung DK, Young WL. Imaging aspirin effect on macrophages in the wall of human cerebral aneurysms using ferumoxytol-enhanced MRI: preliminary results. J Neuroradiol. 2013 Jul;40(3):187-91. doi: 10.1016/j.neurad.2012.09.002. Epub 2013 Feb 18. PMID 23428244